CLINICAL TRIAL: NCT01772472
Title: A Randomized, Multicenter, Open-Label Phase III Study to Evaluate the Efficacy and Safety of Trastuzumab Emtansine Versus Trastuzumab as Adjuvant Therapy for Patients With HER2-Positive Primary Breast Cancer Who Have Residual Tumor Present Pathologically in the Breast or Axillary Lymph Nodes Following Preoperative Therapy
Brief Title: A Study of Trastuzumab Emtansine Versus Trastuzumab as Adjuvant Therapy in Patients With HER2-Positive Breast Cancer Who Have Residual Tumor in the Breast or Axillary Lymph Nodes Following Preoperative Therapy (KATHERINE)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: NSABP Foundation Inc (Network); GBG Forschungs GmbH (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BO27938; 2012-002018-37 (EudraCT Number)
Record Dates: First submitted 2013-01-17; First posted 2013-01-21 (Estimated); Results first posted 2019-10-01 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Trastuzumab; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Trastuzumab (Active Comparator)
  Interventions: Drug: trastuzumab
- Trastuzumab emtansine (Experimental)
  Interventions: Drug: trastuzumab emtansine

INTERVENTIONS:
Drug: trastuzumab — 6 mg/kg intravenously every 3 weeks, 14 cycles
  Arms: Trastuzumab
Drug: trastuzumab emtansine — 3.6 mg/kg intravenously every 3 weeks, 14 cycles
  Arms: Trastuzumab emtansine

SUMMARY:
This 2-arm, randomized, open-label study will evaluate the efficacy and safety of trastuzumab emtansine versus trastuzumab as adjuvant therapy in patients with HER2-positive breast cancer who have residual tumor present in the breast or axillary lymph nodes following preoperative therapy. Eligible patients will be randomized to receive either trastuzumab emtansine 3.6 mg/kg or trastuzumab 6 mg/kg intravenously every 3 weeks for 14 cycles. Radiotherapy and/or hormone therapy will be given in addition if indicated.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient, >/= 18 years of age
* HER2-positive breast cancer
* Histologically confirmed invasive breast carcinoma
* Clinical stage T1-4/N0-3/M0 at presentation (patients with T1a/bN0 tumors will not be eligible)
* Completion of preoperative systemic chemotherapy and HER2-directed treatment consisting of at least 6 cycles of chemotherapy with a total duration of at least 16 weeks, including at least 9 weeks of trastuzumab and at least 9 weeks of taxane-based therapy
* Adequate excision: surgical removal of all clinically evident disease in the breast and lymph nodes as specified in protocol
* Pathological evidence of residual invasive carcinoma in the breast or axillary lymph nodes following completion of preoperative therapy
* An interval of no more than 12 weeks between the date of surgery and the date of randomization
* Known hormone-receptor status
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Adequate hematologic, renal and liver function
* Screening Left ventricular ejection fraction (LVEF) >/= 50% on echocardiogram (ECHO) or multiple-gated acquisition (MUGA) after receiving neoadjuvant chemotherapy and no decrease in LVEF by more than 15% absolute points from the pre-chemotherapy LVEF. Or, if pre-chemotherapy LVEF was not assessed, the screening LVEF must be >/= 55% after completion of neoadjuvant chemotherapy.
* For women who are not postmenopausal or surgically sterile: agreement to remain abstinent or use single or combined contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 7 months after the last dose of study drug
* Documentation of hepatitis B virus and hepatitis C virus serology is required

Exclusion Criteria:

* Stage IV (metastatic) breast cancer
* History of any prior (ipsi- or contralateral breast cancer except lobular carcinoma in situ
* Evidence of clinically evident gross residual or recurrent disease following preoperative therapy and surgery
* Progressive disease during preoperative systemic therapy
* Treatment with any anti-cancer investigational drug within 28 days prior to commencing study treatment
* History of other malignancy within the last 5 years except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, Stage I uterine cancer, or other non-breast malignancies with a similar outcome to those mentioned above
* Patients for whom radiotherapy would be recommended for breast cancer treatment but for whom it is contraindicated because of medical reasons
* Current NCI CTCAE (Version 4.0) Grade >/= 2 peripheral neuropathy
* History of exposure to the following cumulative doses of anthracyclines: Doxorubicin > 240 mg/m2; Epirubicin or Liposomal Doxorubicin-Hydrochloride (Myocet®) > 480 mg/m2; For other anthracyclines, exposure equivalent to doxorubicin > 240 mg/m2
* Cardiopulmonary dysfunction as defined by protocol
* Prior treatment with trastuzumab emtansine
* Current severe, uncontrolled systemic disease
* Pregnant or lactating women
* Any known active liver disease, e.g. due to HBV, HCV, autoimmune hepatic disorders, or sclerosing cholangitis
* Concurrent serious uncontrolled infections requiring treatment or known infection with HIV
* History of intolerance, including Grade 3 to 4 infusion reaction or hypersensitivity to trastuzumab or murine proteins or any components of the product

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1486 (Actual)
Dates: Start 2013-04-03 (Actual); Primary Completion 2018-07-25 (Actual); Study Completion 2024-05-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (268):
- United States (60):
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Todd Cancer Institute at Long Beach Memorial Medical Center, Long Beach, California
  - Chao Family Comprehensive Cancer Center, Orange, California
  - Stanford University Medical Center, Palo Alto, California
  - Kaiser Permanente - San Diego, San Diego, California
  - Breastlink Medical Group Inc, Santa Ana, California
  - Kaiser Permanente - Vallejo, Vallejo, California
  - Kaiser Permanente - Franklin, Denver, Colorado
  - Colorado Cancer Research Program/Admin, Denver, Colorado
  - Yale Cancer Center, New Haven, Connecticut
  - Washington Cancer Institute, Washington D.C., District of Columbia
  - University of Florida, Gainesville, Florida
  - Mount Sinai Medical Center, Miami Beach, Florida
  - UF Health Orlando, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Rush University Medical Center, Chicago, Illinois
  - Edward Cancer Center Naperville, Naperville, Illinois
  - Edward Cancer Center Plainfield, Plainfield, Illinois
  - University of Iowa, Iowa City, Iowa
  - University of Kentucky Medical Center, Lexington, Kentucky
  - Norton Healthcare Inc., Louisville, Kentucky
  - Cancer Care of Maine, Brewer, Maine
  - New England Cancer Specialists, Scarborough, Maine
  - Mercy Medical Center, Baltimore, Maryland
  - Greater Baltimore Medical Center, Baltimore, Maryland
  - Med Star Franklin Square Medical Center/Weinburg Cancer Institute, Baltimore, Maryland
  - Karmanos Cancer Institute, Detroit, Michigan
  - Henry Ford Health System, Detroit, Michigan
  - Spectrum Health Hospitals, Grand Rapids, Michigan
  - Breslin Cancer Center, Lansing, Michigan
  - William Beaumont Hospital, Royal Oak, Michigan
  - US oncology research at Minnesota Oncology, Saint Louis Park, Minnesota
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Sparta Cancer Center, Sparta, New Jersey
  - Columbia University Medical Center, New York, New York
  - Troy Cancer Treatment Program, Troy, New York
  - Carolinas Medical Center, Charlotte, North Carolina
  - Sanford Roger Maris Cancer Center, Fargo, North Dakota
  - Aultman Hospital, Canton, Ohio
  - Fairview Hospital, Cleveland, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Arthur James Cancer Hospital, Columbus, Ohio
  - Columbia River Oncology Program, Portland, Oregon
  - Kimmel Cancer Center Thomas Jefferson University, Philadelphia, Pennsylvania
  - Allegheny Cancer Center, Pittsburgh, Pennsylvania
  - Uni of Pittsburgh, Pittsburgh, Pennsylvania
  - York Hospital, York, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - Baylor College of Medicine, Houston, Texas
  - Houston Methodist Hospital Outpatient Center, Houston, Texas
  - Uni of Texas - Md Anderson Cancer Center, Houston, Texas
  - Joe Arrington Cancer Research & Treatment Center, Lubbock, Texas
  - Hematology Oncology Associates of Fredericksburg, Inc., Fredericksburg, Virginia
  - Centra Alan B. Pearson Regional Cancer Center, Lynchburg, Virginia
  - Virginia Commonwealth University - Massey Cancer Center, Richmond, Virginia
  - Swedish Cancer Institute - Issaquah, Issaquah, Washington
  - Cancer Care Northwest, Spokane, Washington
  - Marshfield Clinic, Marshfield, Wisconsin
- Argentina (3):
  - Fundación CENIT para la Investigación en Neurociencias, Buenos Aires
  - Centro Oncologico Riojano Integral (CORI), La Rioja
  - Instituto de Oncología de Rosario, Rosario
- Austria (3):
  - Tiroler Landeskrankenanstalten Ges.M.B.H., Innsbruck
  - Lkh Salzburg - Univ. Klinikum Salzburg, Salzburg
  - Medizinische Universität Wien, Vienna
- Belgium (4):
  - Cliniques Universitaires St-Luc, Brussels
  - AZ Sint Lucas (Sint Lucas), Ghent
  - CHU de Liège (Sart Tilman), Liège
  - Sint Augustinus Wilrijk, Wilrijk
- Brazil (10):
  - Iop Instituto de Oncologia Do Parana, Curitiba, Paraná
  - UPCO - Unidade de Pesquisas Clínicas em Oncologia, Pelotas, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul
  - Hospital de Cancer de Barretos, Barretos, São Paulo
  - Instituto de Ensino e Pesquisa Sao Lucas - IEP, São Paulo, São Paulo
  - Instituto do Cancer do Estado de Sao Paulo - ICESP, São Paulo, São Paulo
  - Hospital Perola Byington, São Paulo, São Paulo
  - Instituto Nacional de Cancer - INCa, Rio de Janeiro
  - Clinicas Oncologicas Integradas - COI, Rio de Janeiro
- Canada (12):
  - Arthur J.E. Child Comprehensive Cancer Center, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - BC Cancer ? Surrey, Surrey, British Columbia
  - British Columbia Cancer Agency (Bcca) - Vancouver Cancer Centre, Vancouver, British Columbia
  - London Regional Cancer Centre, London, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Princess Margaret Cancer Center, Toronto, Ontario
  - CSSS champlain - Charles-Le Moyne, Greenfield Park, Quebec
  - Centre Hospitalier de l?Université de Montréal (CHUM), Montreal, Quebec
  - Jewish General Hospital, Montreal, Quebec
  - McGill University Health Centre - Glen Site, Montreal, Quebec
  - Hopital du Saint Sacrement, Québec, Quebec
- China (7):
  - the First Hospital of Jilin University, Changchun
  - Sun Yet-sen University Cancer Center, Guangzhou
  - Guangdong General Hospital, Guangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Shandong Cancer Hospital, Jinan
  - Shanghai Jiao Tong University School of Medicine (SJTUSM) - Ruijin Hospital (GuangCi Hospital), Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai
- Colombia (3):
  - Clinica del Country, Bogotá
  - Hospital Pablo Tobon Uribe, Medellin-Antioquia
  - Oncomedica S.A., Montería
- Czechia (3):
  - Fakultni Nemocnice Hradec Kralove, Hradec Králové
  - Fakultni nemocnice Olomouc, Olomouc
  - Vseobecna fakultni nemocnice v Praze, Prague
- France (16):
  - Institut Sainte Catherine, Avignon
  - Hopital Jean Minjoz, Besançon
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Fleyriat, Bourg-en-Bresse
  - Centre Francois Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre de Cancerologie de la Sarthe, Clinique Victor HugoSoReCOH, Le Mans
  - Institut Paoli Calmettes, Marseille
  - Centre Val Aurelle Paul Lamarque, Montpellier
  - Institut Curie, Paris
  - Hopital Saint Louis, Paris
  - Hopital Tenon, Paris
  - Centre Henri Becquerel, Rouen
  - Centre Rene Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Gustave Roussy, Villejuif
- Germany (47):
  - Hämatologie Onkologie im Zentrum MVZ GmbH, Augsburg
  - Onkologische Schwerpunktpraxis Kurfürstendamm, Berlin
  - HELIOS Klinikum Berlin-Buch, Berlin
  - Studienzentrum Berlin City, Berlin
  - Onkologische Schwerpunktpraxis Bielefeld, Bielefeld
  - Klinikum Sindelfingen-Böblingen, Böblingen
  - St. Elisabeth Krankenhaus Köln GmbH, Cologne
  - Kliniken der Stadt Köln gGmbH Krankenhaus Holweide, Cologne
  - St. Johannes-Hospital, Dortmund
  - Luisenkrankenhaus GmbH & Co. KG., Brustzentrum, Düsseldorf
  - Universitätsklinikum Erlangen, Erlangen
  - Universitätsklinikum Essen, Essen
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH, Essen
  - Klinikum Esslingen, Esslingen am Neckar
  - Klinik Johann Wolfgang von Goethe Uni, Frankfurt
  - Hämatologisch-Onkologische Gemeinschaftspraxis am Bethanien-Krankenhaus, Frankfurt am Main
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Evangelische Kliniken Gelsenkirchen GmbH, Gelsenkirchen
  - Universitätsklinikum Greifswald, Greifswald
  - Universitätsklinikum Halle (Saale), Halle
  - Krankenhaus St. Elisabeth und St. Barbara, Klinik für Frauenheilkunde und Geburtshilfe, Halle
  - Kooperatives Mammazentrum Hamburg Krankenhaus Jerusalem, Hamburg
  - St. Barbara-Klinik Hamm-Heessen GmbH, Hamm
  - Diakovere Henriettenstift, Frauenklinik, Hanover
  - Medizinische Hochschule Hannover, Klinik für Frauenheilkunde und Geburtshilfe, Hanover
  - Nationales Centrum für Tumorerkrankungen (NCT), Heidelberg
  - Elisabeth-Krankenhaus Brustzentrum, Kassel
  - Klinikum Kassel GmbH, Kassel
  - UNI-Klinikum Campus Kiel Klinik für Gynäkologie und Geburtshilfe, Kiel
  - Gemeinschaftspraxis für Hämatologie und Onkologie, PD Dr. Bauer, Dr. Thiel, Lebach
  - Praxisklinik Krebsheilkunde für Frauen / Brustzentrum (Dres. Kittel/Klare), Lichtenberg
  - Klinikum der Universität München, München
  - Medizinisches Zentrum für Hämatologie und Onkologie, München
  - MVZ Nordhausen gGmbH, Praxis Dr. Grafe, Nordhausen
  - Sana Klinikum Offenbach GmbH, Offenbach
  - St. Vincenz-Krankenhaus Paderborn, Paderborn
  - Oncologianova GmbH - Gesellschaft für Innovationen in der Onkologie, Recklinghausen
  - Klinikum am Steinenberg Frauenklinik, Reutlingen
  - Universitätsfrauen- und Poliklinik am Klinikum Suedstadt, Rostock
  - Gynäkologie Kompetenzzentrum, Stralsund
  - Robert-Bosch-Krankenhaus, Stuttgart
  - Gemeinschaftspraxis Dr. Kronawitter und Dr. Jung, Traunstein
  - Universitätsklinik Tübingen, Tübingen
  - Universitätsklinikum Ulm Am Michelsberg, Ulm
  - HELIOS Dr. Horst Schmidt Kliniken Wiesbaden, Wiesbaden
  - Marien-Hospital Witten, Witten
  - Hämatologisch-Onkologische Schwerpunktpraxis Dres. Schlag & Schöttker, Würzburg
- Greece (2):
  - Univ General Hosp Heraklion, Heraklion
  - Euromedical General Clinic of Thessaloniki, Thessaloniki
- Guatemala (2):
  - Centro Oncológico Sixtino / Centro Oncológico SA, Guatemala City
  - Grupo Angeles, Guatemala City
- Hong Kong (3):
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
- Ireland (6):
  - Cork Uni Hospital, Cork
  - St Vincent'S Uni Hospital, Dublin
  - Mater Misericordiae Uni Hospital, Dublin
  - Beaumont Hospital, Dublin
  - Galway Uni Hospital, Galway
  - University Hospital Limerick - Oncology, Limerick
- Israel (6):
  - Soroka Medical Center, Beersheba
  - Shaare Zedek Medical Center, Jerusalem
  - Hadassah University Hospital - Ein Kerem, Jerusalem
  - Rabin MC, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Kaplan Medical Center, Rehovot
- Italy (19):
  - Ospedale Antonio Perrino, Brindisi, Apulia
  - Istituto Nazionale Tumori Fondazione G. Pascale, Napoli, Campania
  - Università degli Studi Federico II, Napoli, Campania
  - Policlinico S.Orsola-Malpighi, Bologna, Emilia-Romagna
  - Ausl Di Bologna-Ospedale Bellaria, Bologna, Emilia-Romagna
  - Policlinico Universitario Campus Biomedico, Rome, Lazio
  - Az. Osp. Sant'Andrea, Rome, Lazio
  - IRCCS Istituto Nazionale Per La Ricerca Sul Cancro (IST), Genoa, Liguria
  - Asst Papa Giovanni XXIII, Bergamo, Lombardy
  - Asst Di Cremona, Cremona, Lombardy
  - Irccs Ospedale San Raffaele, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Istituto Europeo Di Oncologia, Milan, Lombardy
  - Asst Di Monza, Monza, Lombardy
  - Fondazione Del Piemonte Per L'oncologia IRCC Di Candiolo, Candiolo, Piedmont
  - Azlenda Ospendaliero-Universitaria Pisana, Pisa, Tuscany
  - Azienda usl 5 Di Pisa-Ospedale Di Pontedera, Pontedera, Tuscany
  - IOV - Istituto Oncologico Veneto - IRCCS, Padua, Veneto
  - A.O.U.I. Verona-Ospedale Borgo Trento, Verona, Veneto
- Mexico (5):
  - Hospital Angeles Metropolitano, Mexico City, Mexico CITY (federal District)
  - Médicos Especialistas en Cáncer SC, Aguascalientes
  - Instituto Nacional de Cancerologia, Distrito Federal
  - Nstituto Nacional de Ciancias Medicas Y Nutricion, Salvador Zubir, Mexico City
  - Oaxaca Site Management Organization, Oaxaca City
- Panama (2):
  - The Panama Clinic, Panama City
  - Centro Oncologico America, Panama City
- Peru (5):
  - Hospital Nacional Carlos Alberto Seguin Escobedo-Essalud, Arequipa
  - Centro Medico Monte Carmelo, Arequipa
  - Hospital IV Alberto Sabogal Sologuren, Bellavista
  - Hospital Nacional Guillermo Almenara Irigoyen, Lima
  - Clinica San Borja, Lima
- Serbia (2):
  - Institute for Oncology and Radiology of Serbia, Belgrade
  - Oncology Institute of Vojvodina, Kamenitz
- South Africa (6):
  - Cape Town Oncology Trials, Cape Town
  - Medical Oncology Centre of Rosebank, Johannesburg
  - Wits Donald Gordon Clinical Trial Centre, Parktown
  - Hopelands Cancer Centre, Pietermaritzburg
  - Cancercare, Port Elizabeth
  - Private Oncology Centre, Pretoria
- Spain (13):
  - Hospital de Donostia, Donostia / San Sebastian, Guipuzcoa
  - Hospital Severo Ochoa, Leganés, Madrid
  - Hospital de Navarra, Navarra, Navarre
  - Complexo Hospitalario de Vigo. Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Hospital Universitari Sant Joan de Reus, Reus, Tarragona
  - Hospital Clínic i Provincial, Barcelona
  - Hospital Universitario La Paz, Madrid
  - Hospital de Madrid Norte Sanchinarro- Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Regional Universitario Carlos Haya, Málaga
  - Hospital Clinico Universitario de Salamanca, Salamanca
  - Hospital Universitario Virgen del Rocio, Seville
  - Instituto Valenciano Oncologia, Valencia
  - Hospital Universitario Dr. Peset, Valencia
- Sweden (3):
  - Gävle Sjukhus, Gävle
  - Skånes University Hospital, Skånes Department of Onclology, Lund
  - Karolinska Hospital, Stockholm
- Switzerland (2):
  - Kantonsspital Aarau AG Medizin Onkologie, Aarau
  - Brust-Zentrum Zürich AG Seefeldstrasse 214 Zürich, Zurich
- Taiwan (5):
  - Taichung Veterans General Hospital, Taichung
  - Veterans General Hospital, Taipei
  - National Taiwan Uni Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Medical Foundation - Linkou, Taoyuan District
- Turkey (Türkiye) (5):
  - Uludag Uni Hospital, Bursa
  - Trakya University Medical Faculty Research And Practice Hospital Medical Oncology Department, Edirne
  - Kartal Dr Lutfi Kirdar Sehir Hastanesi, Istanbul
  - Ege Uni Medical Faculty Hospital, Izmir
  - Inonu University Medical Faculty Turgut Ozal Medical Center Medical Oncology Department, Malatya
- United Kingdom (14):
  - University Hospital Birmingham The Cancer Centre, Queen Elizabeth Hospital, Birmingham
  - Bradford Royal Infirmary, Bradford
  - Bristol Haematology and Oncology centre, Bristol
  - Castle Hill Hospital, Cottingham
  - North Devon District Hospital, Devon
  - Ninewells Hospital, Dundee
  - Huddersfield Royal Infirmary, Huddersfield
  - Leeds Teaching Hosp NHS Trust, Leeds
  - St Thomas Hospital, London
  - Charing Cross Hospital, London
  - Christie Hospital Nhs Trust, Manchester
  - Nottingham City Hospital, Nottingham
  - Weston Park Hospital, Sheffield
  - Royal Cornwall Hospital, Truro

REFERENCES:
- [Derived] Geyer CE Jr, Untch M, Huang CS, Mano MS, Mamounas EP, Wolmark N, Rastogi P, Schneeweiss A, Redondo A, Fischer HH, D'Hondt V, Conlin AK, Guarneri V, Wapnir IL, Jackisch C, Arce-Salinas C, Fasching PA, DiGiovanna MP, Crown JP, Wuelfing P, Shao Z, Rota Caremoli E, Bonnefoi HR, Hennessy BT, Stamatovic L, Castro-Salguero H, Brufsky AM, Knott A, Siddiqui A, Lambertini C, Boulet T, Nyawira B, Restuccia E, Loibl S; KATHERINE Study Group. Survival with Trastuzumab Emtansine in Residual HER2-Positive Breast Cancer. N Engl J Med. 2025 Jan 16;392(3):249-257. doi: 10.1056/NEJMoa2406070. PMID 39813643
- [Derived] von Minckwitz G, Huang CS, Mano MS, Loibl S, Mamounas EP, Untch M, Wolmark N, Rastogi P, Schneeweiss A, Redondo A, Fischer HH, Jacot W, Conlin AK, Arce-Salinas C, Wapnir IL, Jackisch C, DiGiovanna MP, Fasching PA, Crown JP, Wulfing P, Shao Z, Rota Caremoli E, Wu H, Lam LH, Tesarowski D, Smitt M, Douthwaite H, Singel SM, Geyer CE Jr; KATHERINE Investigators. Trastuzumab Emtansine for Residual Invasive HER2-Positive Breast Cancer. N Engl J Med. 2019 Feb 14;380(7):617-628. doi: 10.1056/NEJMoa1814017. Epub 2018 Dec 5. PMID 30516102

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 1486 participants with human epidermal growth factor receptor 2 (HER2)-positive primary breast cancer who had residual invasive disease in either the breast or axillary lymph nodes took part in the study at 268 investigative sites across 28 countries from April 03, 2013 to May 23, 2024.
Pre-assignment Details: Participants received either trastuzumab or trastuzumab emtansine (T-DM1). 1 participant randomized to trastuzumab arm was untreated, later re-randomized to T-DM1 arm & received treatment. Another participant in the trastuzumab arm received 13 cycles of trastuzumab & 1 of T-DM1. Both these participants were included in the trastuzumab ITT population and T-DM1 safety analysis. 1 participant in T-DM1 arm received 9 cycles of trastuzumab & included in trastuzumab safety analysis.
Groups:
- Trastuzumab: Participants received trastuzumab, 6 milligram per kilograms (mg/kg), intravenously (IV), every 3 weeks (Q3W), as a maintenance dose for 14 cycles (1 cycle = 21 days) or until disease recurrence or unacceptable toxicity which ever occurs first.
- Trastuzumab Emtansine: Participants received trastuzumab emtansine, 3.6 mg/kg, IV, Q3W for 14 cycles (1 cycle = 21 days) or until disease recurrence or unacceptable toxicity which ever occurs first.
Period: Overall Study
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Started | 743 | 743
Safety-evaluable (SE) Population (SE population included all randomized participants who received any amount of study treatment.) | 720 (1 participant in trastuzumab emtansine arm received 9 cycles of trastuzumab & included in trastuzumab safety analysis.) | 740 (1 participant randomized to trastuzumab arm was untreated, later re-randomized to trastuzumab emtansine arm & received treatment. Another participant in the trastuzumab arm received 13 cycles of trastuzumab & 1 of trastuzumab emtansine. Both these participants were included in the trastuzumab emtansine safety analysis.)
Completed | 0 | 0
Not Completed | 743 | 743
Not completed — Death | 126 | 94
Not completed — Lost to Follow-up | 51 | 50
Not completed — Other | 9 | 7
Not completed — Physician Decision | 1 | 7
Not completed — Withdrawal by Subject | 115 | 90
Not completed — Follow-up Terminated by Sponsor | 441 | 495

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized to the study regardless of whether they received any study treatment.
Groups:
- Trastuzumab: Participants received trastuzumab, 6 mg/kg, IV, Q3W, as a maintenance dose for 14 cycles (1 cycle = 21 days) or until disease recurrence or unacceptable toxicity which ever occurs first.
- Total: Total of all reporting groups
Arm/Group | Trastuzumab | Trastuzumab Emtansine | Total
Number analyzed (Participants) | 743 | 743 | 1486
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 675 | 685 | 1360
  >=65 years | 68 | 58 | 126
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 740 | 741 | 1481
  Male | 3 | 2 | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 107 | 91 | 198
  Not Hispanic or Latino | 543 | 579 | 1122
  Unknown or Not Reported | 93 | 73 | 166
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 50 | 36 | 86
  Asian | 64 | 65 | 129
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 19 | 21 | 40
  White | 530 | 551 | 1081
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 77 | 69 | 146

OUTCOME MEASURES:

1. Primary Outcome: Invasive Disease-free Survival (IDFS) Rate at 3 Years
Description: IDFS event was defined as the first occurrence of any one of the following events: ipsilateral invasive breast tumor recurrence (i.e., an invasive breast cancer involving the same breast parenchyma as the original primary lesion); ipsilateral local-regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, regional lymph nodes, chest wall and/or skin of the ipsilateral breast); distant recurrence (i.e., evidence of breast cancer in any anatomic site-other than the 2 above-mentioned sites - that has either been histologically confirmed or clinically diagnosed as recurrent invasive breast cancer); contralateral invasive breast cancer; death attributable to any cause including breast cancer, non-breast cancer or unknown cause . 3-year IDFS rate in ITT population was estimated using Kaplan Meier (KM) method and the percentage of participants who were event-free 3 years after randomization was estimated.
Time Frame: At Year 3
Population: ITT population included all participants who were randomized to the study regardless of whether they received any study treatment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 77.12 [73.96 to 80.28] | 88.44 [86.07 to 90.81]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI [0.44 to 0.66]

2. Other Pre Specified Outcome: IDFS Rate at 7 Years
Description: IDFS event was defined as the first occurrence of any one of the following events: ipsilateral invasive breast tumor recurrence (i.e., an invasive breast cancer involving the same breast parenchyma as the original primary lesion); ipsilateral local-regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, regional lymph nodes, chest wall and/or skin of the ipsilateral breast); distant recurrence (i.e., evidence of breast cancer in any anatomic site-other than the 2 above-mentioned sites - that has either been histologically confirmed or clinically diagnosed as recurrent invasive breast cancer); contralateral invasive breast cancer; death attributable to any cause including breast cancer, non-breast cancer or unknown cause . 7-year IDFS rate in ITT population was estimated using KM method and the percentage of participants who were event-free 7 years after randomization was estimated.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 67.11 [63.53 to 70.68] | 80.82 [77.86 to 83.78]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI [0.44 to 0.66]

3. Other Pre Specified Outcome: IDFS Rate at 8 Years
Description: IDFS event was defined as the first occurrence of any one of the following events: ipsilateral invasive breast tumor recurrence (i.e., an invasive breast cancer involving the same breast parenchyma as the original primary lesion); ipsilateral local-regional invasive breast cancer recurrence (i.e., an invasive breast cancer in the axilla, regional lymph nodes, chest wall and/or skin of the ipsilateral breast); distant recurrence (i.e., evidence of breast cancer in any anatomic site-other than the 2 above-mentioned sites - that has either been histologically confirmed or clinically diagnosed as recurrent invasive breast cancer); contralateral invasive breast cancer; death attributable to any cause including breast cancer, non-breast cancer or unknown cause . 8-year IDFS rate in ITT population was estimated using KM method and the percentage of participants who were event-free 8 years after randomization was estimated.
Time Frame: At Year 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 64.57 [60.90 to 68.23] | 79.11 [76.03 to 82.19]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.54, 95% CI 2-sided [0.44 to 0.66]

4. Secondary Outcome: IDFS Including Second Primary Non-breast Cancer (SPNBC) Rate at 3 Years
Description: IDFS including SPNBC was defined the same way as IDFS but including second primary non breast invasive cancer as an event (with the exception of non-melanoma skin cancers and carcinoma in situ [CIS] of any site). IDFS event was defined as outlined in the description for IDFS rate outcome measure (OM) number 1. 3-year IDFS including SPNBC rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 3 years after randomization was estimated.
Time Frame: At Year 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 76.98 [73.82 to 80.15] | 87.87 [85.45 to 90.29]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.46 to 0.69]

5. Secondary Outcome: IDFS Including SPNBC Rate at 7 Years
Description: IDFS including SPNBC was defined the same way as IDFS but including second primary non breast invasive cancer as an event (with the exception of non-melanoma skin cancers and CIS of any site). IDFS event was defined as outlined in the description for IDFS rate OM number 1. 7-year IDFS including SPNBC rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 7 years after randomization was estimated.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 66.19 [62.59 to 69.80] | 79.81 [76.79 to 82.82]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI [0.46 to 0.69]

6. Secondary Outcome: IDFS Including SPNBC Rate at 8 Years
Description: IDFS including SPNBC was defined the same way as IDFS but including second primary non breast invasive cancer as an event (with the exception of non-melanoma skin cancers and CIS of any site). IDFS event was defined as outlined in the description for IDFS rate OM number 1. 8-year IDFS including SPNBC rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 8 years after randomization was estimated.
Time Frame: At Year 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 63.65 [59.96 to 67.34] | 77.76 [74.60 to 80.92]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.57, 95% CI 2-sided [0.46 to 0.69]

7. Secondary Outcome: Disease-free Survival (DFS) Rate at 3 Years
Description: DFS was defined as the time between randomization and the date of the first occurrence of an IDFS event including SPNBC event or contralateral or ipsilateral ductal carcinoma in situ (DCIS). IDFS event was defined as outlined in the description for IDFS rate OM number 1. 3-year DFS rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 3 years after randomization was estimated.
Time Frame: At Year 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 76.98 [73.82 to 80.15] | 87.59 [85.15 to 90.03]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI [0.48 to 0.70]

8. Secondary Outcome: DFS Rate at 7 Years
Description: DFS was defined as the time between randomization and the date of the first occurrence of an IDFS event including SPNBC event or contralateral or ipsilateral DCIS. IDFS event was defined as outlined in the description for IDFS rate OM number 1. 7-year DFS rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 7 years after randomization was estimated.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 66.03 [62.42 to 69.64] | 79.37 [76.33 to 82.42]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI [0.48 to 0.70]

9. Secondary Outcome: DFS Rate at 8 Years
Description: DFS was defined as the time between randomization and the date of the first occurrence of an IDFS event including SPNBC event or contralateral or ipsilateral DCIS. IDFS event was defined as outlined in the description for IDFS rate OM number 1. 8-year DFS rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 8 years after randomization was estimated.
Time Frame: At Year 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 63.49 [59.80 to 67.18] | 77.14 [73.95 to 80.33]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.58, 95% CI 2-sided [0.48 to 0.70]

10. Secondary Outcome: Overall Survival (OS) Rate at 5 Years
Description: OS was defined as the time from randomization to death due to any cause. 5-year OS event-free rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 5 years after randomization was estimated.
Time Frame: At Year 5
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 87.71 [85.20 to 90.22] | 91.40 [89.30 to 93.50]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p = 0.0082, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.53 to 0.91]

11. Secondary Outcome: OS Rate at 7 Years
Description: OS was defined as the time from randomization to death due to any cause. 7-year OS event-free rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 7 years after randomization was estimated.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 84.38 [81.59 to 87.17] | 89.07 [86.72 to 91.43]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p = 0.0082, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI [0.53 to 0.91]

12. Secondary Outcome: OS Rate at 8 Years
Description: OS was defined as the time from randomization to death due to any cause. 8-year OS event-free rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 8 years after randomization was estimated.
Time Frame: At Year 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 81.91 [78.94 to 84.89] | 87.16 [84.62 to 89.70]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p = 0.0082, Log Rank; Hazard Ratio (HR) = 0.70, 95% CI 2-sided [0.53 to 0.91]

13. Secondary Outcome: Distant Recurrence-free Interval (DRFI) Rate at 3 Years
Description: DRFI was defined as the time between randomization and the date of distant breast cancer recurrence. 3-year DRFI event-free rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 3 years after randomization was estimated.
Time Frame: At Year 3
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 83.26 [80.43 to 86.08] | 89.95 [87.72 to 92.19]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI [0.47 to 0.76]

14. Secondary Outcome: DRFI Rate at 7 Years
Description: DRFI was defined as the time between randomization and the date of distant breast cancer recurrence. 7-year DRFI event-free rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 7 years after randomization was estimated.
Time Frame: At Year 7
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 76.22 [72.95 to 79.48] | 84.55 [81.82 to 87.27]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI [0.47 to 0.76]

15. Secondary Outcome: DRFI Rate at 8 Years
Description: DRFI was defined as the time between randomization and the date of distant breast cancer recurrence. 8-year DRFI event-free rate in the ITT population was estimated using KM method, and the percentage of participants who were event-free 8 years after randomization was estimated.
Time Frame: At Year 8
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
percentage of participants | 74.28 [70.90 to 77.65] | 83.82 [81.03 to 86.62]
Statistical Analysis 1: Comparison: Trastuzumab vs Trastuzumab Emtansine; Test type: Superiority; p < .0001, Log Rank; Hazard Ratio (HR) = 0.60, 95% CI 2-sided [0.47 to 0.76]

16. Secondary Outcome: Percentage of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: AE=any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. AE can therefore be any unfavorable & unintended sign (including abnormal laboratory finding), symptom/disease temporally associated with use of a medicinal product, whether or not considered related to medicinal product. SAE=any AE that met any given criteria: fatal (i.e. AE causes/leads to death); life-threatening (i.e. AE, in view of investigator, placed the participant at immediate risk of death); required/prolonged inpatient hospitalization; resulted in persistent or significant disability/incapacity (i.e. AE results in substantial disruption of participant's ability to conduct normal life functions); congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug; significant medical event in investigator's judgment. Percentages have been rounded off.
Time Frame: From signing of informed consent till end of follow up (up to approximately 131 months)
Population: SE population included all randomized participants who received any amount of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 720 | 740
percentage of participants
  AEs | 93.3 | 98.8
  SAEs | 8.1 | 12.7

17. Secondary Outcome: Percentage of Participants With Cardiac Events as Adjudicated by the Cardiac Review Committee
Description: Cardiac events were defined as death from cardiac cause or severe congestive heart failure (New York Heart Association [NYHA] Class III or IV) with a decrease in left ventricular ejection fraction (LVEF) of 10 percentage points or more from baseline to an LVEF of < 50%. Other cardiac-related events (e.g., any symptomatic congestive heart failure [CHF] associated with a 10% drop in LVEF to < 50%; asymptomatic declines in LVEF requiring dose delay) were summarized as adjudicated by the Cardiac Review Committee. Percentages have been rounded off.
Time Frame: Up to approximately 126 months
Population: SE population included all randomized participants who received any amount of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 720 | 740
percentage of participants | 4.2 | 3.1

18. Secondary Outcome: Percentage of Participants With Hepatotoxicity Events as Adjudicated by the Hepatic Review Committee
Description: Hepatotoxicity events were summarized by treatment arm. Hepatotoxicity events were assessed using liver function laboratory test (LFT) results which included the analysis of baseline and post-baseline levels of alanine transaminase (ALT), aspartate aminotransferase (AST), total bilirubin (TBILI), and alkaline phosphatase (ALK). Hepatic events, as adjudicated by the Hepatic Review Committee, are summarized. Percentages have been rounded off.
Time Frame: Up to approximately 64 months
Population: SE population included all randomized participants who received any amount of study treatment.
Measure: Number; unit: percentage of participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 720 | 740
percentage of participants | 0.1 | 0.5

19. Secondary Outcome: Number of Participants Who Discontinued Treatment Due to AEs
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. Participants were treated for up to 14 cycles (1 cycle = 21 days).
Time Frame: Up to approximately 9.6 months
Population: SE population included all randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 720 | 740
Participants | 15 | 134

20. Secondary Outcome: Number of Participants With AEs and SAEs Leading to Death
Description: An AE was any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of causal attribution. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. A SAE was any AE that met any of the following criteria: fatal (i.e., the AE actually causes or leads to death); life-threatening (i.e., the AE, in the view of the investigator, placed the participant at immediate risk of death); required or prolonged inpatient hospitalization; resulted in persistent or significant disability/incapacity (i.e., the AE results in substantial disruption of the participant's ability to conduct normal life functions); congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug; significant medical event in the investigator's judgment.
Time Frame: From signing of informed consent till end of follow up (up to approximately 131 months)
Population: SE population included all randomized participants who received any amount of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 720 | 740
Participants | 0 | 1

21. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire - Core 30 (QLQ-C30)
Description: The EORTC QLQ-C30 consists of 30 questions which assess five functional domains (physical, role, cognitive, emotional, and social), a global health status/quality of life (GHS/QoL) scale, three symptom scales (fatigue, pain, nausea, and vomiting), five single items (dyspnea, appetite loss, sleep disturbance, constipation, and diarrhea), and a perceived financial impact of the disease item. Most questions used a 4-point scale (1= Not at all to 4 = Very much; 2 questions used a 7-point scale [1 = very poor to 7 = Excellent]). Obtained scores are linearly transformed to a score range of 0-100, whereby higher scores indicate greater functioning, greater quality of life, or a greater degree of symptoms. A positive change from baseline indicates improvement.
Time Frame: Baseline, Cycles 5 &11, Follow-up (FU) Month 6, FU Month 12 (1 cycle = 21 days)
Population: ITT population included all participants who were randomized to the study regardless of whether they received any study treatment. Overall number analyzed is the number of participants with data available for analysis. Number analyzed per timepoint are unique number of participants out of all the assessed participants with data available for analysis at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
score on a scale
  Baseline: Appetite Loss: number analyzed (Participants) | 624 | 645
  Baseline: Appetite Loss | 7.9 (17.4) | 7.1 (16.4)
  Change at Cycle 5: Appetite Loss: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Appetite Loss | 1.0 (18.7) | 6.5 (23.7)
  Change at Cycle 11: Appetite Loss: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Appetite Loss | -0.5 (17.2) | 2.9 (20.2)
  Change at FU Month 6: Appetite Loss: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Appetite Loss | -1.6 (18.3) | -1.7 (19.9)
  Change at FU Month 12: Appetite Loss: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Appetite Loss | 0.5 (20.3) | -1.9 (20.1)
  Baseline: Constipation: number analyzed (Participants) | 624 | 645
  Baseline: Constipation | 9.8 (20.2) | 9.5 (19.0)
  Change at Cycle 5: Constipation: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Constipation | 1.0 (22.4) | 4.6 (22.6)
  Change at Cycle 11: Constipation: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Constipation | 3.4 (23.6) | 7.3 (23.1)
  Change at FU Month 6: Constipation: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Constipation | 4.1 (23.7) | 3.7 (23.3)
  Change at FU Month 12: Constipation: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Constipation | 3.2 (23.2) | 4.3 (24.6)
  Baseline: Diarrhea: number analyzed (Participants) | 624 | 645
  Baseline: Diarrhea | 8.8 (17.6) | 6.4 (14.9)
  Change at Cycle 5: Diarrhea: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Diarrhea | -1.6 (19.3) | -1.5 (19.5)
  Change at Cycle 11: Diarrhea: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Diarrhea | -0.4 (21.4) | -2.4 (17.5)
  Change at FU Month 6: Diarrhea: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Diarrhea | -3.4 (18.5) | -1.9 (18.3)
  Change at FU Month 12: Diarrhea: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Diarrhea | -2.8 (18.9) | -1.6 (18.4)
  Baseline: Dyspnea: number analyzed (Participants) | 624 | 645
  Baseline: Dyspnea | 12.7 (20.7) | 11.0 (18.8)
  Change at Cycle 5: Dyspnea: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Dyspnea | 2.3 (21.9) | 4.1 (22.4)
  Change at Cycle 11: Dyspnea: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Dyspnea | 2.8 (21.2) | 2.7 (20.4)
  Change at FU Month 6: Dyspnea: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Dyspnea | 3.3 (22.8) | 3.8 (22.7)
  Change at FU Month 12: Dyspnea: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Dyspnea | 3.9 (24.9) | 5.3 (22.4)
  Baseline: Fatigue: number analyzed (Participants) | 624 | 645
  Baseline: Fatigue | 29.2 (21.1) | 28.0 (20.0)
  Change at Cycle 5: Fatigue: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Fatigue | 1.1 (20.1) | 5.5 (19.7)
  Change at Cycle 11: Fatigue: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Fatigue | 1.1 (20.5) | 3.8 (21.3)
  Change at FU Month 6: Fatigue: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Fatigue | -1.4 (21.9) | -0.1 (22.2)
  Change at FU Month 12: Fatigue: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Fatigue | -0.1 (23.3) | -0.1 (22.1)
  Baseline: Financial Difficulties: number analyzed (Participants) | 604 | 635
  Baseline: Financial Difficulties | 28.6 (33.3) | 27.6 (31.9)
  Change at Cycle 5: Financial Difficulties: number analyzed (Participants) | 530 | 548
  Change at Cycle 5: Financial Difficulties | -3.1 (26.5) | -3.0 (28.0)
  Change at Cycle 11: Financial Difficulties: number analyzed (Participants) | 472 | 480
  Change at Cycle 11: Financial Difficulties | -5.1 (27.6) | -1.7 (28.7)
  Change at FU Month 6: Financial Difficulties: number analyzed (Participants) | 393 | 444
  Change at FU Month 6: Financial Difficulties | -8.4 (28.3) | -6.5 (30.6)
  Change at FU Month 12: Financial Difficulties: number analyzed (Participants) | 367 | 413
  Change at FU Month 12: Financial Difficulties | -10.9 (30.5) | -7.3 (31.0)
  Baseline: Insomnia: number analyzed (Participants) | 624 | 645
  Baseline: Insomnia | 30.6 (30.8) | 30.6 (29.2)
  Change at Cycle 5: Insomnia: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Insomnia | 1.9 (28.4) | 1.3 (29.7)
  Change at Cycle 11: Insomnia: number analyzed (Participants) | 494 | 494
  Change at Cycle 11: Insomnia | 2.4 (29.9) | 1.5 (30.3)
  Change at FU Month 6: Insomnia: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Insomnia | 1.8 (31.3) | -0.9 (32.1)
  Change at FU Month 12: Insomnia: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Insomnia | 0.3 (30.4) | 0.7 (31.7)
  Baseline: Nausea/Vomiting: number analyzed (Participants) | 624 | 645
  Baseline: Nausea/Vomiting | 3.3 (9.0) | 2.8 (8.0)
  Change at Cycle 5: Nausea/Vomiting: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Nausea/Vomiting | 1.5 (11.2) | 3.2 (12.5)
  Change at Cycle 11: Nausea/Vomiting: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Nausea/Vomiting | 1.3 (12.8) | 3.0 (11.8)
  Change at FU Month 6: Nausea/Vomiting: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Nausea/Vomiting | 0.8 (10.4) | 0.2 (11.1)
  Change at FU Month 12: Nausea/Vomiting: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Nausea/Vomiting | 0.4 (10.5) | 1.2 (10.9)
  Baseline: Pain: number analyzed (Participants) | 624 | 645
  Baseline: Pain | 22.2 (22.2) | 22.6 (22.8)
  Change at Cycle 5: Pain: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Pain | 0.0 (23.2) | 1.8 (23.9)
  Change at Cycle 11: Pain: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Pain | 0.1 (23.1) | 2.1 (24.4)
  Change at FU Month 6: Pain: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Pain | -0.3 (24.6) | -0.5 (24.3)
  Change at FU Month 12: Pain: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Pain | -1.2 (25.6) | -0.8 (25.4)
  Baseline: Cognitive Functioning: number analyzed (Participants) | 624 | 645
  Baseline: Cognitive Functioning | 83.3 (20.2) | 84.4 (19.0)
  Change at Cycle 5: Cognitive Functioning: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Cognitive Functioning | -3.8 (18.4) | -4.5 (18.7)
  Change at Cycle 11: Cognitive Functioning: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Cognitive Functioning | -5.4 (21.3) | -5.3 (19.6)
  Change at FU Month 6: Cognitive Functioning: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Cognitive Functioning | -4.1 (22.0) | -6.1 (21.6)
  Change at FU Month 12: Cognitive Functioning: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Cognitive Functioning | -4.9 (22.2) | -6.9 (21.7)
  Baseline: Emotional Functioning: number analyzed (Participants) | 624 | 645
  Baseline: Emotional Functioning | 75.0 (22.0) | 75.2 (21.2)
  Change at Cycle 5: Emotional Functioning: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Emotional Functioning | -0.4 (20.0) | -1.3 (21.3)
  Change at Cycle 11: Emotional Functioning: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Emotional Functioning | -1.0 (21.3) | 0.1 (22.0)
  Change at FU Month 6: Emotional Functioning: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Emotional Functioning | -2.9 (22.0) | -0.8 (23.3)
  Change at FU Month 12: Emotional Functioning: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Emotional Functioning | -2.0 (22.7) | -1.6 (23.5)
  Baseline: Physical Functioning: number analyzed (Participants) | 624 | 645
  Baseline: Physical Functioning | 84.5 (15.3) | 85.8 (14.1)
  Change at Cycle 5: Physical Functioning: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Physical Functioning | 0.3 (12.9) | -1.6 (12.7)
  Change at Cycle 11: Physical Functioning: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Physical Functioning | 1.9 (14.2) | -0.6 (14.6)
  Change at FU Month 6: Physical Functioning: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Physical Functioning | 2.8 (15.4) | 0.7 (15.1)
  Change at FU Month 12: Physical Functioning: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Physical Functioning | 2.7 (14.5) | 0.8 (14.5)
  Baseline: Role Functioning: number analyzed (Participants) | 624 | 645
  Baseline: Role Functioning | 77.5 (25.0) | 78.6 (23.3)
  Change at Cycle 5: Role Functioning: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Role Functioning | 2.0 (24.3) | -0.2 (24.1)
  Change at Cycle 11: Role Functioning: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Role Functioning | 4.0 (24.3) | 0.6 (24.5)
  Change at FU Month 6: Role Functioning: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Role Functioning | 7.4 (25.8) | 3.6 (26.7)
  Change at FU Month 12: Role Functioning: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Role Functioning | 8.0 (27.5) | 4.6 (25.5)
  Baseline: Social Functioning: number analyzed (Participants) | 624 | 645
  Baseline: Social Functioning | 77.1 (24.1) | 76.8 (23.2)
  Change at Cycle 5: Social Functioning: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Social Functioning | 4.0 (22.5) | 1.6 (23.8)
  Change at Cycle 11: Social Functioning: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Social Functioning | 5.8 (24.0) | 2.5 (23.6)
  Change at FU Month 6: Social Functioning: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Social Functioning | 8.5 (23.7) | 6.5 (26.1)
  Change at FU Month 12: Social Functioning: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Social Functioning | 9.5 (25.1) | 7.4 (26.4)
  Baseline: Global Health Status: number analyzed (Participants) | 624 | 645
  Baseline: Global Health Status | 71.2 (19.3) | 71.4 (18.0)
  Change at Cycle 5: Global Health Status: number analyzed (Participants) | 558 | 571
  Change at Cycle 5: Global Health Status | 0.6 (18.9) | -1.9 (19.6)
  Change at Cycle 11: Global Health Status: number analyzed (Participants) | 496 | 496
  Change at Cycle 11: Global Health Status | 1.7 (17.8) | -0.5 (19.9)
  Change at FU Month 6: Global Health Status: number analyzed (Participants) | 410 | 462
  Change at FU Month 6: Global Health Status | 2.5 (19.3) | 2.0 (19.2)
  Change at FU Month 12: Global Health Status: number analyzed (Participants) | 384 | 430
  Change at FU Month 12: Global Health Status | 3.2 (19.5) | 2.8 (20.1)

22. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire - Breast Cancer (QLQ-BR23)
Description: EORTC-QLQ-BR23 is a 23-item breast cancer-specific companion module to the EORTC-QLQ-C30 and consists of four functional scales (body image, sexual enjoyment, sexual functioning, future perspective [FP]) and four symptom scales (systemic side effects [SE], upset by hair loss, arm symptoms, breast symptoms). Questions used 4-point scale (1=not at all, 2=a little, 3=quite a bit, 4=very much). Obtained scores are linearly transformed to a score range of 0-100. High score for functional scale indicated high/better level of functioning/healthy functioning. Higher scores for symptom scales represent higher levels of symptoms/problems. For functional scales, positive change from baseline indicated deterioration in QOL and negative change from baseline indicated an improvement in QOL. For symptom scales, positive change from baseline indicated an improvement in QOL and negative change from baseline indicated a deterioration in QOL.
Time Frame: Baseline, Cycles 5 &11, Follow-up (FU) Month 6, FU Month 12 (1 cycle = 21 days)
Population: as for outcome 21
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Trastuzumab | Trastuzumab Emtansine
Number analyzed (Participants) | 743 | 743
score on a scale
  Baseline: Body Image: number analyzed (Participants) | 622 | 645
  Baseline: Body Image | 69.8 (28.5) | 67.5 (28.5)
  Change at Cycle 5: Body Image: number analyzed (Participants) | 555 | 571
  Change at Cycle 5: Body Image | 1.5 (20.5) | 4.6 (22.7)
  Change at Cycle 11: Body Image: number analyzed (Participants) | 493 | 495
  Change at Cycle 11: Body Image | 3.4 (24.4) | 5.7 (23.9)
  Change at FU Month 6: Body Image: number analyzed (Participants) | 409 | 462
  Change at FU Month 6: Body Image | 3.6 (25.1) | 7.8 (25.8)
  Change at FU Month 12: Body Image: number analyzed (Participants) | 383 | 428
  Change at FU Month 12: Body Image | 6.2 (27.1) | 6.1 (27.2)
  Baseline: FP: number analyzed (Participants) | 622 | 645
  Baseline: FP | 51.3 (31.2) | 50.1 (31.7)
  Change at Cycle 5: FP: number analyzed (Participants) | 555 | 571
  Change at Cycle 5: FP | 2.6 (28.3) | 6.5 (29.9)
  Change at Cycle 11: FP: number analyzed (Participants) | 493 | 495
  Change at Cycle 11: FP | 6.3 (30.0) | 6.1 (31.4)
  Change at FU Month 6: FP: number analyzed (Participants) | 409 | 462
  Change at FU Month 6: FP | 7.7 (33.5) | 8.1 (34.6)
  Change at FU Month 12: FP: number analyzed (Participants) | 383 | 428
  Change at FU Month 12: FP | 8.1 (31.1) | 8.2 (33.0)
  Baseline: Sexual Enjoyment: number analyzed (Participants) | 218 | 241
  Baseline: Sexual Enjoyment | 50.9 (28.8) | 52.3 (28.5)
  Change at Cycle 5: Sexual Enjoyment: number analyzed (Participants) | 147 | 172
  Change at Cycle 5: Sexual Enjoyment | 2.3 (26.4) | -1.9 (24.6)
  Change at Cycle 11: Sexual Enjoyment: number analyzed (Participants) | 128 | 137
  Change at Cycle 11: Sexual Enjoyment | 4.4 (27.5) | 4.4 (24.5)
  Change at FU Month 6: Sexual Enjoyment: number analyzed (Participants) | 104 | 126
  Change at FU Month 6: Sexual Enjoyment | 3.2 (28.1) | 0.3 (27.5)
  Change at FU Month 12: Sexual Enjoyment: number analyzed (Participants) | 95 | 114
  Change at FU Month 12: Sexual Enjoyment | 5.6 (26.0) | 1.8 (26.2)
  Baseline: Sexual Function: number analyzed (Participants) | 550 | 564
  Baseline: Sexual Function | 20.2 (23.6) | 22.0 (23.4)
  Change at Cycle 5: Sexual Function: number analyzed (Participants) | 456 | 466
  Change at Cycle 5: Sexual Function | 3.3 (20.0) | 2.3 (20.0)
  Change at Cycle 11: Sexual Function: number analyzed (Participants) | 393 | 382
  Change at Cycle 11: Sexual Function | 3.1 (20.8) | 1.9 (20.3)
  Change at FU Month 6: Sexual Function: number analyzed (Participants) | 321 | 360
  Change at FU Month 6: Sexual Function | 5.1 (23.9) | 4.3 (23.1)
  Change at FU Month 12: Sexual Function: number analyzed (Participants) | 289 | 319
  Change at FU Month 12: Sexual Function | 5.9 (23.7) | 5.2 (22.7)
  Baseline: Arm Symptoms: number analyzed (Participants) | 622 | 645
  Baseline: Arm Symptoms | 24.6 (21.1) | 24.5 (21.0)
  Change at Cycle 5: Arm Symptoms: number analyzed (Participants) | 555 | 571
  Change at Cycle 5: Arm Symptoms | -2.8 (20.9) | -2.6 (23.0)
  Change at Cycle 11: Arm Symptoms: number analyzed (Participants) | 493 | 495
  Change at Cycle 11: Arm Symptoms | -2.6 (21.2) | 0.2 (24.2)
  Change at FU Month 6: Arm Symptoms: number analyzed (Participants) | 409 | 462
  Change at FU Month 6: Arm Symptoms | -3.0 (23.5) | -1.3 (24.2)
  Change at FU Month 12: Arm Symptoms: number analyzed (Participants) | 383 | 428
  Change at FU Month 12: Arm Symptoms | -5.7 (22.8) | -1.5 (22.6)
  Baseline: Breast Symptoms: number analyzed (Participants) | 622 | 645
  Baseline: Breast Symptoms | 22.7 (19.1) | 21.4 (17.9)
  Change at Cycle 5: Breast Symptoms: number analyzed (Participants) | 555 | 571
  Change at Cycle 5: Breast Symptoms | -1.1 (20.3) | -1.1 (19.1)
  Change at Cycle 11: Breast Symptoms: number analyzed (Participants) | 493 | 495
  Change at Cycle 11: Breast Symptoms | -3.7 (19.8) | -0.6 (19.5)
  Change at FU Month 6: Breast Function: number analyzed (Participants) | 409 | 462
  Change at FU Month 6: Breast Function | -6.5 (20.0) | -2.2 (19.7)
  Change at Follow-up Month 12: Breast Function: number analyzed (Participants) | 383 | 428
  Change at Follow-up Month 12: Breast Function | -8.3 (19.9) | -3.8 (19.2)
  Baseline: Systemic Therapy Side Effects (SE): number analyzed (Participants) | 622 | 645
  Baseline: Systemic Therapy Side Effects (SE) | 16.7 (13.7) | 16.9 (14.1)
  Change at Cycle 5: Systemic Therapy SE: number analyzed (Participants) | 555 | 571
  Change at Cycle 5: Systemic Therapy SE | 0.7 (13.0) | 5.5 (15.3)
  Change at Cycle 11: Systemic Therapy SE: number analyzed (Participants) | 493 | 495
  Change at Cycle 11: Systemic Therapy SE | 1.2 (12.2) | 4.2 (15.4)
  Change at FU Month 6: Systemic Therapy SE: number analyzed (Participants) | 409 | 462
  Change at FU Month 6: Systemic Therapy SE | 1.9 (13.9) | 1.1 (15.3)
  Change at FU Month 12: Systemic Therapy SE: number analyzed (Participants) | 383 | 428
  Change at FU Month 12: Systemic Therapy SE | 1.3 (13.9) | 1.4 (16.3)
  Baseline: Upset by Hair Loss Item: number analyzed (Participants) | 77 | 96
  Baseline: Upset by Hair Loss Item | 40.3 (35.6) | 50.7 (38.4)
  Change at Cycle 5: Upset by Hair Loss Item: number analyzed (Participants) | 13 | 17
  Change at Cycle 5: Upset by Hair Loss Item | -5.1 (38.1) | -17.6 (39.3)
  Change at Cycle 11: Upset by Hair Loss Item: number analyzed (Participants) | 14 | 14
  Change at Cycle 11: Upset by Hair Loss Item | -28.6 (45.0) | -14.3 (33.9)
  Change at FU Month 6: Upset by Hair Loss Item: number analyzed (Participants) | 25 | 22
  Change at FU Month 6: Upset by Hair Loss Item | -12.0 (47.0) | -15.2 (42.1)
  Change at FU Month 12: Upset by Hair Loss Item: number analyzed (Participants) | 23 | 21
  Change at FU Month 12: Upset by Hair Loss Item | -2.9 (37.5) | -14.3 (41.6)

23. Secondary Outcome: Serum Concentrations of Trastuzumab Emtansine
Time Frame: Pre-infusion on Cycles 1, 2, 4 and 5; 15-30 minutes and 2 hours post-infusion on Cycles 1 and 4; treatment discontinuation/completion visit (up to approximately 64 months) (1 cycle = 21 days)
Population: Pharmacokinetic (PK)-evaluable population included all participants who received at least 1 dose of trastuzumab emtansine and had at least one evaluable post dose PK sample. Overall number analyzed is the number of participants with data available for analysis. Number analyzed per timepoint are unique number of participants out of all the assessed participants with data available for analysis at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (ug/mL)
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 423
micrograms per milliliter (ug/mL)
  Pre-infusion on Cycle 1: number analyzed (Participants) | 406
  Pre-infusion on Cycle 1 | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable as the samples were below the limit of quantification. The samples were taken prior to administration of the first dose.
  15-30 minutes post-infusion on Cycle 1: number analyzed (Participants) | 402
  15-30 minutes post-infusion on Cycle 1 | 63.0 (101.8)
  2 hours post-infusion on Cycle 1: number analyzed (Participants) | 388
  2 hours post-infusion on Cycle 1 | 67.4 (60.0)
  Pre-infusion on Cycle 2: number analyzed (Participants) | 383
  Pre-infusion on Cycle 2 | 1.69 (110.7)
  Pre-infusion on Cycle 4: number analyzed (Participants) | 379
  Pre-infusion on Cycle 4 | 1.73 (95.7)
  15-30 minutes post-infusion on Cycle 4: number analyzed (Participants) | 375
  15-30 minutes post-infusion on Cycle 4 | 68.5 (59.4)
  2 hours post-infusion on Cycle 4: number analyzed (Participants) | 358
  2 hours post-infusion on Cycle 4 | 66.4 (71.0)
  Pre-infusion on Cycle 5: number analyzed (Participants) | 336
  Pre-infusion on Cycle 5 | 1.67 (99.3)
  Treatment Completion/Discontinuation: number analyzed (Participants) | 323
  Treatment Completion/Discontinuation | 0.323 (265.3)

24. Secondary Outcome: Plasma Concentrations of Deacetyl Mercapto 1-Oxopropyl Maytansine (DM1)
Description: Concentration of DM1 in plasma was measured through the samples obtained from participants randomized to the trastuzumab emtansine arm. DM1 is an ant-microtubule agent derived from maytansine. In transtuzumab entansine, DM1 is linked to the antibody transtuzumab thus helping the drug to specifically target the HER 2- positive cancer cells.
Time Frame: Pre-infusion, 15-30 minutes and 2 hour post-infusion on Cycles 1 and 4 (1 cycle = 21 days)
Population: PK-evaluable population included all participants who received atleast 1 dose of trastuzumab emtansine and had at least one evaluable post dose PK sample. Overall number analyzed is the number of participants with data available for analysis. Number analyzed per timepoint are unique number of participants out of all the assessed participants with data available for analysis at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 417
nanograms per milliliter (ng/mL)
  Pre-infusion on Cycle 1: number analyzed (Participants) | 401
  Pre-infusion on Cycle 1 | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable as majority of the values were lower than reportable.
  15-30 minutes post-infusion on Cycle 1: number analyzed (Participants) | 397
  15-30 minutes post-infusion on Cycle 1 | 4.21 (57.4)
  2 hours post-infusion on Cycle 1: number analyzed (Participants) | 387
  2 hours post-infusion on Cycle 1 | 3.44 (38.2)
  Pre-infusion on Cycle 4: number analyzed (Participants) | 361
  Pre-infusion on Cycle 4 | 0.372 (NA) — The geometric coefficient of variation was not estimable as majority of the values were lower than reportable or zero.
  15-30 minutes post-infusion on Cycle 4: number analyzed (Participants) | 359
  15-30 minutes post-infusion on Cycle 4 | 4.81 (48.8)
  2 hours post-infusion on Cycle 4: number analyzed (Participants) | 347
  2 hours post-infusion on Cycle 4 | 3.70 (41.0)

25. Secondary Outcome: Serum Concentrations of Trastuzumab
Time Frame: Pre-infusion and 15-30 minutes post-infusion on Cycles 1 and 4; Treatment completion/discontinuation visit (up to approximately 64 months) (1 cycle = 21 days)
Population: PK-evaluable population included all participants who received at least 1 dose of trastuzumab and had at least one evaluable post dose PK sample. Overall number analyzed is the number of participants with data available for analysis. Number analyzed per timepoint are unique number of participants out of all the assessed participants with data available for analysis at the specified timepoint. Different participants may have contributed data for each timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Trastuzumab
Number analyzed (Participants) | 404
ug/mL
  Pre-infusion on Cycle 1: number analyzed (Participants) | 388
  Pre-infusion on Cycle 1 | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable as the samples were below the limit of quantification. The samples were taken prior to administration of the first dose.
  15-30 minutes post-infusion on Cycle 1: number analyzed (Participants) | 384
  15-30 minutes post-infusion on Cycle 1 | 208 (43.1)
  Pre-infusion on Cycle 4: number analyzed (Participants) | 361
  Pre-infusion on Cycle 4 | 64.8 (60.6)
  15-30 minutes post-infusion on Cycle 4: number analyzed (Participants) | 355
  15-30 minutes post-infusion on Cycle 4 | 218 (47.2)
  Treatment Completion/Discontinuation: number analyzed (Participants) | 325
  Treatment Completion/Discontinuation | 58.7 (86.3)

26. Secondary Outcome: Serum Concentrations of Total Trastuzumab
Description: Total trastuzumab is the sum of conjugated and unconjugated trastuzumab. Blood and serum samples were obtained from participants randomized to the trastuzumab arm.
Time Frame: Pre-infusion on Day 1 of Cycles 1, 2, 4, and 5; 15-30 minutes and 2 hours post-infusion on Day 1 of Cycles 1 and 4 (1 cycle = 21 days)
Population: as for outcome 25
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ug/mL
Arm/Group | Trastuzumab
Number analyzed (Participants) | 421
ug/mL
  Pre-infusion on Cycle 1: number analyzed (Participants) | 390
  Pre-infusion on Cycle 1 | NA (NA) — The geometric mean and geometric coefficient of variation were not estimable as the samples were below the limit of quantification. The samples were taken prior to administration of the first dose.
  15-30 minutes post-infusion on Cycle 1: number analyzed (Participants) | 418
  15-30 minutes post-infusion on Cycle 1 | 71.8 (154.7)
  2 hours post-infusion on Cycle 1: number analyzed (Participants) | 50
  2 hours post-infusion on Cycle 1 | 81.4 (74.3)
  Pre-infusion on Cycle 2: number analyzed (Participants) | 42
  Pre-infusion on Cycle 2 | 7.93 (256.8)
  Pre-infusion on Cycle 4: number analyzed (Participants) | 391
  Pre-infusion on Cycle 4 | 13.7 (78.0)
  15-30 minutes post-infusion on Cycle 4: number analyzed (Participants) | 361
  15-30 minutes post-infusion on Cycle 4 | 76.9 (46.5)
  2 hours post-infusion on Cycle 4: number analyzed (Participants) | 37
  2 hours post-infusion on Cycle 4 | 81.5 (34.0)
  Pre-infusion on Cycle 5: number analyzed (Participants) | 31
  Pre-infusion on Cycle 5 | 8.90 (125.0)

27. Secondary Outcome: Median Duration of Trastuzumab Emtansine Exposure
Description: Treatment duration was defined as the time between the first and the last infusion of trastuzumab emtansine.
Time Frame: Up to 12 months
Population: SE population included all randomized participants who received any amount of study treatment.
Measure: Median (Full Range); unit: months
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 740
months | 10 [1 to 12]

28. Secondary Outcome: Number of Participants With Positive Anti-drug Antibodies (ADAs) to Trastuzumab Emtansine
Description: ADA-positive participants after drug administration were determined for participants exposed to trastuzumab emtansine. For determining post-baseline incidence, participants were considered to be ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following study drug exposure, or if they were ADA-positive at baseline and the titer of 1 or more post-baseline samples was at least 0.60 titer units (t.u.) greater than the baseline titer result. The total number of participants who developed ADAs to trastuzumab emtansine was determined by summing the ADA-positive participants across all timepoints.
Time Frame: Baseline (Day1 of Cycle1) and Post Baseline (Day 1 of Cycle 4 up to 3-4 months after last dose of the drug [up to approximately 13.6 months])
Population: SE Population included all randomized participants who received any amount of study treatment. Overall number analyzed is the number of participants with data available for analysis. Number analyzed is the number of participants with data available for analysis at the specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab Emtansine
Number analyzed (Participants) | 740
Participants
  Baseline: number analyzed (Participants) | 410
  Baseline | 17
  Post-baseline: number analyzed (Participants) | 401
  Post-baseline | 16

29. Secondary Outcome: Number of Participants With Positive ADAs to Trastuzumab
Description: ADA-positive participants after drug administration were determined for participants exposed to trastuzumab. For determining post-baseline incidence, participants were considered to be ADA-positive if they were ADA-negative or had missing data at baseline but developed an ADA response following study drug exposure, or if they were ADA-positive at baseline and the titer of 1 or more post-baseline samples was at least 0.60 t.u. greater than the baseline titer result. The total number of participants who developed ADAs to trastuzumab was determined by summing the ADA-positive participants across all timepoints.
Time Frame: as for outcome 28
Population: as for outcome 28
Measure: Count of Participants; unit: Participants
Arm/Group | Trastuzumab
Number analyzed (Participants) | 720
Participants
  Baseline: number analyzed (Participants) | 386
  Baseline | 11
  Post-baseline: number analyzed (Participants) | 392
  Post-baseline | 15

ADVERSE EVENTS:
Time Frame: From signing of informed consent till the end of follow-up (up to approximately 131 months)
Description: AE(s): SE Population. All-cause mortality: ITT population.1 participant randomized to trastuzumab arm was untreated, later re-randomized to T-DM1 arm & received treatment. Another participant in trastuzumab arm received 13 cycles of trastuzumab & 1 of T-DM1. Both these participants were included in the trastuzumab ITT population & T-DM1 safety analysis (SA). 1 participant in T-DM1 arm received 9 cycles of trastuzumab & included in trastuzumab SA.
Arm/Group | Trastuzumab | Trastuzumab Emtansine
All-Cause Mortality (participants affected / at risk) | 126/743 | 94/743
Serious Adverse Events (participants affected / at risk) | 58/720 | 94/740
Other Adverse Events (participants affected / at risk) | 633/720 | 719/740
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab (N=720) | Trastuzumab Emtansine (N=740)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 3 (3) | 2 (2)
CARDIOGENIC SHOCK (Cardiac disorders) | 1 (1) | 0 (0)
PERICARDITIS (Cardiac disorders) | 1 (1) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (2) | 3 (3)
COLITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 1 (1) | 1 (1)
HAEMORRHOIDS (Gastrointestinal disorders) | 1 (1) | 0 (0)
ILEAL PERFORATION (Gastrointestinal disorders) | 0 (0) | 1 (1)
IMPAIRED GASTRIC EMPTYING (Gastrointestinal disorders) | 0 (0) | 1 (1)
LARGE INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 1 (1)
PANCREATITIS (Gastrointestinal disorders) | 1 (1) | 0 (0)
VOMITING (Gastrointestinal disorders) | 2 (3) | 3 (4)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 3 (3)
PYREXIA (General disorders) | 0 (0) | 1 (1)
SYSTEMIC INFLAMMATORY RESPONSE SYNDROME (General disorders) | 1 (1) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 1 (1) | 1 (1)
GALLBLADDER POLYP (Hepatobiliary disorders) | 1 (1) | 0 (0)
HEPATIC CYST (Hepatobiliary disorders) | 0 (0) | 1 (1)
HEPATITIS (Hepatobiliary disorders) | 0 (0) | 1 (1)
NODULAR REGENERATIVE HYPERPLASIA (Hepatobiliary disorders) | 0 (0) | 2 (2)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 4 (4)
ABSCESS INTESTINAL (Infections and infestations) | 0 (0) | 1 (1)
APPENDICITIS (Infections and infestations) | 0 (0) | 2 (2)
BRONCHITIS (Infections and infestations) | 1 (1) | 3 (3)
CELLULITIS (Infections and infestations) | 2 (2) | 1 (1)
CYSTITIS (Infections and infestations) | 1 (1) | 0 (0)
DEVICE RELATED INFECTION (Infections and infestations) | 0 (0) | 5 (5)
DIVERTICULITIS (Infections and infestations) | 0 (0) | 1 (1)
ENTEROCOLITIS INFECTIOUS (Infections and infestations) | 1 (1) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 2 (2)
IMPLANT SITE CELLULITIS (Infections and infestations) | 1 (1) | 0 (0)
INFECTED SEROMA (Infections and infestations) | 0 (0) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 1 (1)
MASTITIS (Infections and infestations) | 6 (7) | 8 (8)
PERIRECTAL ABSCESS (Infections and infestations) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 2 (2) | 6 (6)
SKIN INFECTION (Infections and infestations) | 1 (1) | 2 (2)
STAPHYLOCOCCAL BACTERAEMIA (Infections and infestations) | 0 (0) | 1 (1)
TONSILLITIS (Infections and infestations) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 1 (1)
VASCULAR DEVICE INFECTION (Infections and infestations) | 0 (0) | 1 (1)
VESTIBULAR NEURONITIS (Infections and infestations) | 1 (1) | 0 (0)
VULVITIS (Infections and infestations) | 0 (0) | 1 (1)
WOUND INFECTION (Infections and infestations) | 2 (2) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
POST PROCEDURAL HAEMORRHAGE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
RADIATION PNEUMONITIS (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
RADIUS FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
SEROMA (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
TIBIA FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
ULNA FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND COMPLICATION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
WOUND DEHISCENCE (Injury, poisoning and procedural complications) | 1 (1) | 3 (3)
WRIST FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1)
EJECTION FRACTION DECREASED (Investigations) | 1 (1) | 0 (0)
PLATELET COUNT DECREASED (Investigations) | 0 (0) | 10 (10)
TROPONIN T INCREASED (Investigations) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
COLON CANCER STAGE I (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
ENDOMETRIAL ADENOCARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
INTRADUCTAL PROLIFERATIVE BREAST LESION (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
PITUITARY TUMOUR BENIGN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 0 (0) | 1 (1)
HAEMORRHAGE INTRACRANIAL (Nervous system disorders) | 0 (0) | 1 (1)
NEURALGIA (Nervous system disorders) | 0 (0) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 3 (3)
SYNCOPE (Nervous system disorders) | 0 (0) | 2 (2)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (2)
SUICIDAL IDEATION (Psychiatric disorders) | 0 (0) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 1 (1)
BLADDER PAIN (Renal and urinary disorders) | 1 (1) | 0 (0)
HEAVY MENSTRUAL BLEEDING (Reproductive system and breast disorders) | 0 (0) | 1 (1)
OVARIAN CYST (Reproductive system and breast disorders) | 1 (1) | 0 (0)
UTERINE HAEMORRHAGE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
UTERINE OBSTRUCTION (Reproductive system and breast disorders) | 1 (1) | 0 (0)
UTERINE PROLAPSE (Reproductive system and breast disorders) | 1 (1) | 0 (0)
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
PULMONARY FIBROSIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
TELANGIECTASIA (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
EMBOLISM (Vascular disorders) | 3 (3) | 1 (1)
HAEMATOMA (Vascular disorders) | 1 (1) | 0 (0)
HYPERTENSION (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Trastuzumab (N=720) | Trastuzumab Emtansine (N=740)
ANAEMIA (Blood and lymphatic system disorders) | 60 (79) | 74 (90)
LACRIMATION INCREASED (Eye disorders) | 13 (13) | 41 (44)
ABDOMINAL PAIN (Gastrointestinal disorders) | 42 (49) | 55 (66)
CONSTIPATION (Gastrointestinal disorders) | 59 (66) | 125 (151)
DIARRHOEA (Gastrointestinal disorders) | 89 (116) | 91 (117)
DRY MOUTH (Gastrointestinal disorders) | 9 (9) | 100 (109)
NAUSEA (Gastrointestinal disorders) | 93 (111) | 308 (441)
STOMATITIS (Gastrointestinal disorders) | 25 (28) | 80 (96)
VOMITING (Gastrointestinal disorders) | 37 (45) | 107 (140)
CHILLS (General disorders) | 14 (16) | 39 (57)
FATIGUE (General disorders) | 243 (276) | 363 (456)
INFLUENZA LIKE ILLNESS (General disorders) | 86 (96) | 100 (138)
OEDEMA PERIPHERAL (General disorders) | 52 (56) | 29 (33)
PAIN (General disorders) | 92 (113) | 90 (107)
PYREXIA (General disorders) | 29 (32) | 76 (98)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 53 (65) | 59 (70)
URINARY TRACT INFECTION (Infections and infestations) | 37 (39) | 64 (79)
RADIATION SKIN INJURY (Injury, poisoning and procedural complications) | 199 (207) | 186 (196)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 41 (51) | 172 (209)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 40 (44) | 210 (255)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 13 (14) | 61 (68)
BLOOD BILIRUBIN INCREASED (Investigations) | 2 (2) | 49 (74)
NEUTROPHIL COUNT DECREASED (Investigations) | 36 (47) | 61 (78)
PLATELET COUNT DECREASED (Investigations) | 17 (21) | 206 (261)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 41 (61) | 61 (82)
DECREASED APPETITE (Metabolism and nutrition disorders) | 16 (19) | 65 (74)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 14 (20) | 48 (61)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 158 (175) | 202 (233)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 66 (73) | 53 (57)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 35 (38) | 51 (54)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 45 (45) | 33 (36)
MYALGIA (Musculoskeletal and connective tissue disorders) | 80 (87) | 113 (126)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 71 (82) | 87 (99)
DIZZINESS (Nervous system disorders) | 57 (61) | 69 (77)
DYSGEUSIA (Nervous system disorders) | 11 (12) | 57 (58)
HEADACHE (Nervous system disorders) | 124 (148) | 209 (289)
PARAESTHESIA (Nervous system disorders) | 40 (43) | 56 (68)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 50 (51) | 136 (146)
ANXIETY (Psychiatric disorders) | 42 (44) | 27 (29)
DEPRESSION (Psychiatric disorders) | 44 (47) | 41 (44)
INSOMNIA (Psychiatric disorders) | 86 (95) | 101 (110)
BREAST PAIN (Reproductive system and breast disorders) | 41 (49) | 52 (55)
COUGH (Respiratory, thoracic and mediastinal disorders) | 86 (93) | 100 (112)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 52 (57) | 62 (69)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 25 (30) | 158 (225)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 33 (36) | 37 (39)
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 21 (23) | 39 (44)
DRY SKIN (Skin and subcutaneous tissue disorders) | 36 (40) | 48 (52)
PRURITUS (Skin and subcutaneous tissue disorders) | 42 (44) | 52 (58)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 26 (27) | 43 (50)
HOT FLUSH (Vascular disorders) | 144 (152) | 94 (98)
HYPERTENSION (Vascular disorders) | 34 (38) | 42 (59)
LYMPHOEDEMA (Vascular disorders) | 48 (51) | 36 (36)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT01772472/Prot_002.pdf
  • Statistical Analysis Plan (2023-06-20): https://cdn.clinicaltrials.gov/large-docs/72/NCT01772472/SAP_003.pdf